CLINICAL TRIAL: NCT02076880
Title: Investigation of Endocrin-metabolic Modifications Related to Diabetes Improvement After Sleeve Gastrectomy in Severly Obese
Brief Title: SLEEVEDIAB To Explore the Early and Late Metabolic Effects of Sleeve Gastrectomy in Obese Patients
Acronym: SLEEVEDIAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 9016; 2012-A00962-41 (Other: ID-RCB - ANSM)
Record Dates: First submitted 2013-12-17; First posted 2014-03-04 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2013-09

CONDITIONS: Severe Obesity; Type 2 Diabetes
Keywords: Type 2 diabetes; Obesity; Sleeve gastrectomy; Insulin; GLP-1
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2; Obesity; Insulin Resistance | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm with caloric restriction (Experimental): Patients in this arm will have, during 7 days before surgery, a caloric restriction of 1000 kcal per day compared to the usual food intake. They will be hospitalized during this period.
  Intervention: caloric restriction
  Interventions: Other: Caloric restriction
- Arm without caloric restriction (Experimental): Patients in this arm will not have a caloric restriction before surgery.
  Intervention: No caloric restriction
  Interventions: Other: No caloric restriction

INTERVENTIONS:
Other: Caloric restriction — Caloric restriction of 1000 kcal per day compared to the usual food intake.
  * usual breakfast of the patient (possibly limited in quantity)
  * midday and evening meals from mixed and dehydrated meals, soups with protein and dairy desserts sweetened
  Arms: Arm with caloric restriction
Other: No caloric restriction — No change in eating habits to patients in this arm
  Arms: Arm without caloric restriction

SUMMARY:
Sleeve gastrectomy is a restrictive procedure based on the removal of a large part of the gastric fundus. According to a recent randomized study, weight loss and resolution of diabetes are comparable to that obtained after gastric by-pass (79.7 % versus 80.3%), but with a lower morbidity. The mechanisms involved in the rapid resolution of diabetes after sleeve gastrectomy remain poorly understood, as no specific study in patients with type 2 diabetic obese are available. An increase in post- absorptive levels of Glucagon-like Peptide 1(GLP-1), Peptide YY(PYY) and insulin has been reported, but in non-diabetic subjects mostly. The important caloric restriction in the early postoperative period indeed improves hepatic insulin resistance, regardless of weight loss. Specific metabolic and hormonal effects of this surgical procedure cannot be excluded.The aim of our study is to explore the early and late metabolic effects of sleeve gastrectomy in severely obese patients with non-insulin-treated type 2 diabetes. We will also evaluate insulin sensitivity, insulin secretion and incretin effect. We will include 14 obese patients with type 2 diabetes, considered eligible to bariatric surgery according to HAS criteria, and whose diabetes treatment involves only metformin, sulfonylurea and glinides. They will be randomized to a 1-week caloric restriction period or no caloric restriction, immediately before surgery. Test meals with dosages of blood glucose, insulin, C-peptide, adiponectin, leptin, GLP-1, PYY and ghrelin will be performed before and after caloric restriction, and 1 week, 3 month, 6 month and 12 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* Age between 18-65 years (inclusive)
* Men or women receiving effective contraception, postmenopausal or sterile
* type 2 diabetes treated with no drugs or oral anti-diabetic agents metformin, sulfonylurea or glinides
* Body mass index 35 kg / m² or above
* eligible to bariatric surgery according to HAS criteria

Exclusion Criteria:

* Treatment of diabetes with GLP1 analogues, DPP-IV (dipeptidyl-peptidase IV) or insulin
* Treatment with drugs that modify glucose homeostasis: glucocorticoids, anorexigens, antihistaminics, psychotropic drugs especially serotonergic antidepressants (except for the occasional use of a hypnotic or anxiolytic), atropine, laxatives, thyroid hormones (with the exception of a substitution dose ensuring a stable euthyroid at baseline), beta blockers, diuretics
* Pregnancy, intention of being pregnant, breastfeeding.
* Inability to understand the nature and aims of the study or to communicate with the investigator- High probability of non
* compliance with the protocol
* Simultaneous participation in another trial
* No affiliation to the French social security
* Loss of personal capacity resulting in state protection
* Deprivation of liberty by judicial or administrative decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change of area under the curve of post prandial glycemia | Baseline to day 7 after surgery

SECONDARY OUTCOMES:
Change in insulin sensitivity, Change in insulin secretion, Change in incretins | Blood samples at D-15, D-7 before surgery, D7, D80, D170, D350 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Florence GALTIER, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHU Montpellier, Montpellier, France